CLINICAL TRIAL: NCT06695455
Title: The Effect of an Auditory Rhythmic Cue on the Frequency of Rolling in Patients with Dysphagia and Parkinson's Disease: a Pilot Study
Brief Title: The Effect of an Auditory Rhythmic Cue on the Frequency of Rolling in Patients with Dysphagia and Parkinson's Disease
Acronym: Rhythm'nRoll
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital La Musse (Other)
Collaborators: France Parkinson Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A02487-38
Record Dates: First submitted 2024-11-14; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Oral Festination; Lingual Pumping; Dysphagia; Swallowing Disorder; PARKINSON DISEASE (Disorder)
Keywords: oral festination; lingual pumping; dysphagia; swallowing disorder; parkinson disease; rhythmic auditory cue; rehabilitation; behavioral intervention
MeSH Terms: conditions — Deglutition Disorders; Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Interventional research with minimal risks and constraints Prospective, Interventional, Monocentric, without a control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental arm - dysphagic parkinson patient (Experimental): dysphagic parkinson patient
  Interventions: Behavioral: Swallowing rehabilitation by rhythmic auditory cue

INTERVENTIONS:
Behavioral: Swallowing rehabilitation by rhythmic auditory cue — Three assessments, each spread over two days, will be administered at three different time points during the study: before the experiment (T0), after 7 weeks of the experiment (T1), and 3 months after the intervention (T2). The evaluation will include a pharyngography as well as a clinical assessment of swallowing and rhythmic abilities.
  Each subject will be invited to participate in 3 individual rehabilitation sessions per week for 7 weeks, conducted by a speech therapist at La Musse Hospital. Each session will be structured similarly: the subject will be asked to swallow their saliva, followed by a nectar-like texture (IDDSI 2) and a pudding-like texture (IDDSI 4), timed to the rhythm of a metronome. The rhythm will vary throughout the sessions. The goal will be to get as close as possible to the rhythm of a healthy swallow.

SUMMARY:
The main objective of this clinical study is to measure the effect of rhythmic auditory cueing, introduced in rehabilitation with three weekly sessions over a period of 7 weeks, on the frequency of rolling in idiopathic Parkinson's disease patients using pharyngography (swallowing radiography). The primary question of this study is:

Does the rhythmic cueing introduced in rehabilitation significantly reduce the frequency of rolling in dysphagic Parkinson's patients?

The researchers will assess the various stages of swallowing before, after, and 3 months after the rehabilitation protocol, focusing on the oral phase to determine if rhythmic auditory cueing reduces the frequency of rolling.

Participants will be required to:

* Perform three complete assessments (clinical speech therapy examination + pharyngography) before the protocol, after the protocol, and 3 months post-protocol.
* Attend three times per week for 7 weeks at the La Musse hospital to participate in the protocol sessions under the supervision of a speech therapist.

DETAILED DESCRIPTION:
Dysphagia can negatively affect the quality of life of patients. Indeed, it leads to difficulties during oral intake (food, drinks, and medications), weight loss, dehydration, malnutrition, and limitations in social activities. Depression is frequently associated with a reduced quality of life in Parkinson's patients with swallowing disorders. Additionally, aspiration pneumonia due to aspiration events is one of the main causes of hospitalization in Parkinson's patients, and it can lead to severe complications and sometimes death.

This clinical study focuses on "rolling," also known as oropharyngeal festination, which is an involuntary, repetitive, anteroposterior movement of the tongue at the level of the soft palate, performed before the food bolus is swallowed.

Rolling is an intrinsically rhythmic movement. The few studies conducted on the subject agree, however, that freezing of gait (difficulties in initiating movement, stopping in front of an obstacle, or navigating around it) and rolling share common pathophysiological mechanisms. Freezing of gait is not limited to a deficit within the locomotor network but rather reflects a more general deficit affecting spatiotemporal coordination across various tasks, just like rolling.

The use of rhythmic auditory cueing (applying rhythmic auditory training to intrinsically rhythmic movements, such as walking, with the aim of achieving more functional movement patterns) has been evaluated in different studies and has proven effective in reducing the frequency of freezing of gait in Parkinson's patients. It thus seems relevant to apply this rehabilitation method to rolling in these same patients to study the effect of auditory cueing on rolling. The secondary objectives will mainly focus on evaluating the effect of auditory cueing on the swallowing abilities of Parkinson's patients, their physical health, and their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease established by a neurologist using a DAT SCAN and clinical examination;
* Presence of a swallowing disorder, specifically rolling;
* Patient affiliated with the social security system;
* Patient aged 18 years or older

Exclusion Criteria:

* Severe pharyngeal dysphagia (leading to aspiration with nectar and pudding textures);
* Severe cognitive impairment (score <24 on the Mini Mental Parkinson test);
* Known deafness/profound hearing loss;
* Patients under legal protection measures;
* History of reconstructive ENT surgery at the oropharyngeal level;
* Neurological history that could cause a swallowing disorder (e.g., stroke);
* Patient with a gastrostomy and no oral feeding;
* Ongoing speech therapy for swallowing;
* The patient is included in another research protocol;
* Pregnant women or women suspected of being pregnant;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-09-05 (Estimated)

PRIMARY OUTCOMES:
The measurement of the frequency of rolling per minute during a pharyngography | Pre-test (before the rehabilitation protocol), Post-test (after the rehabilitation protocol), and Follow-up test (3 months after the completion of the protocol).
  Multiple measurements will be taken to calculate the average.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital La Musse - La Renaissance Sanitaire, Saint-Sébastien-de-Morsent, Normandy, France

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF